CLINICAL TRIAL: NCT01668342
Title: Mobile Phone Text Message Program to Understand Symptoms and Improve Outcomes in Minor Head Injury Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO12030542
Record Dates: First submitted 2012-07-10; First posted 2012-08-20 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Head Injury, Minor
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS assessments & feedback (Experimental): Daily symptom assessments of headaches, trouble ocncentrating and irritability/anxiety with self-care feedback based on response severity.
  Interventions: Behavioral: SMS assessments & feedback
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: SMS assessments & feedback — Daily symptom assessments tied to tailored feedback
  Arms: SMS assessments & feedback

SUMMARY:
Mild traumatic brain injury (MTBI) is frequently seen in the ED, post-concussive symptoms are common post-injury, and few MTBI patients receive treatment or follow-up for these symptoms. Cell phones are ubiquitous, text messaging (SMS) is a cheap and increasingly common form of communication, potentially allowing for accurate assessment of symptom patterns after MTBI and provision of basic education support . The investigators seek to assess the feasibility of using SMS to collect symptoms related to MTBI in patients either discharged from the ED or admitted to the inpatient trauma unit. The investigators also seek to explore how SMS-based symptom reports correlate with phone-based follow-up reports at 14 days and whether additional SMS-based educational feedback alters daily symptom patterns.

DETAILED DESCRIPTION:
The investigators seek to assess the feasibility of using SMS to collect symptoms related to MTBI in patients either discharged from the ED or admitted to the inpatient trauma unit. The investigators also seek to explore how SMS-based symptom reports correlate with phone-based follow-up reports at 14 days and whether additional SMS-based educational feedback alters daily symptom patterns at 3-months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of minor traumatic brain injury
* English speaking
* Owns a cell phone with SMS

Exclusion Criteria:

* Critically ill

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Rivermead Post Concussive Questionnaire | 14 days

SECONDARY OUTCOMES:
Rivermead Post Concussive Questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Suffoletto, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center-Mercy Hospital, Pittsburgh, Pennsylvania, United States